CLINICAL TRIAL: NCT05400915
Title: Two-Part, Phase Ib/II, Open Label, Single-Arm, Multi-center Study to Evaluate the Safety and Efficacy of Varlitinib in Combination With Weekly Paclitaxel in EGFR/HER2 Co-expressing Advanced or Metastatic Gastric Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-1011
Record Dates: First submitted 2022-05-18; First posted 2022-06-02 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer
Keywords: EGFR/HER2 Co-expressing gastric cancer; Varlitinib
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Variltinib, Paclitaxel (Experimental)
  Interventions: Drug: Variltinib, Paclitaxel

INTERVENTIONS:
Drug: Variltinib, Paclitaxel — Varlitinib will be administered orally to the study participants at doses 300mg, BID in combination with the weekly intravenous infusion of Paclitaxel for 3 weeks with a rest period of 1 week.

SUMMARY:
Phase Ib part of this study determines the recommended phase II dose schedule based on ASLAN001-004 phase Ib (dose-confirmation study of Varlitinib combined with weekly paclitaxel and carboplatin or trastuzumab (Herceptin) in advanced solid tumours). Phase II part of this study further assesses the safety and clinical efficacy of this combination treatment as a second line treatment in EGFR/HER2 co-expressing advanced or metastatic gastric cancer.

DETAILED DESCRIPTION:
This is a two-part, Phase Ib/II, Open label, single arm, multicenter study to determine the maximum tolerated dose (MTD) and the recommended dose schedule of varlitinib in combination with paclitaxel and to further ASLAN001-017_Clinical Study Protocol Version 01_09 Oct 2018 CONFIDENTIAL 7 assess the safety and clinical efficacy of this combined treatment in EGFR/HER2 co-expressing advanced or metastatic gastric cancer after first line treatment. The objective of this trial is to allow development of an effective chemotherapeutic regimen in patients with advanced/metastatic gastric cancer with EGFR/HER-2 co-expression. This trial will also be included in second line Umbrella trial in Yonsei Cancer Center (YCC) (Figure 1).

Patients with EGFR and HER2 co-expression will be confirmed by immunohistochemistry (IHC) and NGS in a central laboratory (Yonsei Cancer Center), and those who meet all eligibility criteria will be enrolled in this study. The patients enrolled in the study will receive combined treatment with varlitinib and paclitaxel until progressive disease is confirmed or at least 1 discontinuation criterion is met (i.e development of intolerable toxicities, patient"s refusal or consent withdrawal or death). Based on previously reported study results, we arrived at an assumption that about 20-25% of screened patients will be categorized as EGFR and HER2 co-expressing gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding and complying with the requirements of the study and have signed the Informed Consent Form (ICF).
2. Able to communicate well with the Investigator and understand and comply with the requirements of the study.
3. Has a histologically or cytologically confirmed diagnosis of advanced or metastatic gastric adenocarcinoma (systemic metastasis or locally advanced unresectable gastric cancer). A subject must have previously received 1st line chemotherapy including fluoropyrimidine and/or platinum and have showed progression.
4. Not received paclitaxel-based chemotherapy previously.
5. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or1
6. Has a measurable or evaluable disease as determined by RECIST 1.1 criteria.
7. Able to swallow orally administered medication.
8. Life expectancy of at least 3 months
9. Has an adequate baseline organ function defined as:

   * White blood cells ≥3000/mm3 and neutrophils ≥1500/mm3
   * Platelets ≥100000/mm3
   * Hemoglobin ≥9.0 g/dL
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 × upper limit of normal (ULN) of the study site (or ≤5.0 × ULN in patients with liver metastases)
   * Total bilirubin ≤2.0 × ULN
   * Creatinine≤1.5 × ULN or creatinine clearance (either measured value or estimated value using the Cockcroft-Gault equation) >60ml/min.

Part 1, Phase Ib

11.Subjects will be included regardless of EGFR and HER-2 Status

Part 2, Phase II

12. Provision of an unstained, archived tumor tissue sample in a quantity sufficient to allow for central analysis of EGFR and HER2 expression status.

13. Tumours with immunohistochemistry (IHC) evidence of expression of HER1 (at level of +, or ++, or +++) and HER-2 (at level of +, or ++, or +++) using standard criteria. Also, Subjects with HER-2 IHC (at level of +, or ++, or +++) and EGFR gene amplification/ mutation by NGS are included.

Exclusion Criteria:

1. Has multiple cancers (with the exception of completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, and superficial bladder cancer, and any other cancers that have not recurred for at least 5 years)
2. Has a current or past history of interstitial lung disease or pulmonary fibrosis diagnosed on imaging (preferably CT) or clinical findings
3. Has brain or leptomeningeal metastases. Patients may be randomized for the study if they are asymptomatic and require no treatment.
4. History of uncontrollable or significant cardiovascular disease meeting any of the following;

   * myocardial infarction within 180 days before study enrolment
   * uncontrolled angina pectoris within 180 days before study enrolment
   * New York Heart Association (NYHA) Class III or IV congestive heart failure
   * uncontrolled hypertension despite appropriate treatment (e.g., systolic blood pressure ≥150mmHg or diastolic blood pressure ≥90 mmHg lasting 24 hours or more)
   * arrhythmia requiring treatment
   * baseline corrected QT interval (Fridericia"s formula) (QTcF) > 450 ms or patients with known long QT syndrome; torsade de pointes
5. Has an active systemic infection requiring treatment.
6. Has a contraindication to paclitaxel.
7. Has undergone surgery (any surgery involving general anesthesia) within 28 days before study treatment.
8. Subjects with malabsorption syndrome, diseases significantly affecting gastrointestinal function, has total gastrectomy, or difficulty in swallowing and retaining oral medications.
9. Has received radiotherapy for gastric cancer within 28 days before treatment or radiotherapy for bone metastases within 14 days before treatment
10. Positive test result for human immunodeficiency virus-1 (HIV-1) antibody, Hepatitis B surface protein (HBs) antigen and HBV titer>2000 IU/ml (10,000 copy/ml), or hepatitis C virus (HCV) antibody positive result
11. Any unresolved Grade 2 (per CTCAE v4.0) toxicity from previous anti-cancer therapy at the time of enrollment such as neuropathy, except alopecia or anemia
12. Previously treated with varlitinib
13. Unable to comply to the study protocol
14. Have participated in a study involving another investigational drug within 21 days prior to the first dose of study drug
15. Has a history of drug hypersensitivity reactions or hypersensitivity to drugs chemically related to the study drug.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
(Phase Ib) Maximum Tolerated dose | 3 years
(Phase Ib) Dose limiting Toxicity | 3 years
(Phase II) Progression-free survival | 3 years
  Progression-free survival (PFS): Defined as the time from start of study treatment until the date of objective disease progression or death (by any cause in the absence of disease progression) Progression is defined in accordance with the RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Overall Survival | 3 years
  Overall Survival (OS): Defined as the time from start of study treatment until death by any cause. Any subject not known to have died at the time of the analysis will be censored based on the last recorded date on which the subject was known to be alive.
Objective Response Rate | 3 years
  Objective Response Rate (ORR)- Objective response rate is defined as the number (%) of patients with at least one confirmed visit response of CR or PR.
Disease Control Rate | 3 years
  Disease Control Rate (DCR): Defined as the proportion of subjects with a best objective response (BOR) of complete response (CR) or partial response (PR), or stable disease maintained for a minimum of twelve weeks (± 5 days) from start of treatment, as defined by the RECIST v1.1 criteria.
Progression-free survival | 3 years
  Progression-free survival (PFS): Defined as the time from start of study treatment until the date of objective disease progression or death (by any cause in the absence of disease progression) Progression is defined in accordance with the RECIST v1.1 criteria. Determination of PFS rate at 24 weeks.
Number of Participants With Adverse Events That Are Related to Treatment | 3 years
  Safety and tolerability of the Varlitinib and Paclitaxel combination therapy as determined by adverse events categorized in accordance with CTCAE 4.03 Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: SUN YOUNG RHA, Principal Investigator — Yonsei Cancer Center, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Yonsei Cancer Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No